CLINICAL TRIAL: NCT01367340
Title: Effect of Physical Activity Intervention on Mobility Changes and Participation for School-Age Children With Spastic Diplegia and After Resistance Training
Brief Title: Effect of Physical Activity Intervention Children With Spastic Diplegia After Resistance Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0993702914; 98-2314-B-002-011-MY3 (Other Grant/Funding Number: NSC of ROC)
Record Dates: First submitted 2010-08-09; First posted 2011-06-07 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-02

CONDITIONS: Cerebral Palsy; Spastic Diplegia
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise and physical activity (Experimental)
  Interventions: Behavioral: Loaded sit-to-stand resistance exercise; Behavioral: Physical activity intervention
- Exercise only (Active Comparator)
  Interventions: Behavioral: Loaded sit-to-stand resistance exercise

INTERVENTIONS:
Behavioral: Loaded sit-to-stand resistance exercise — Loaded STS exercise at home, 3 times a week for 6 weeks
Behavioral: Physical activity intervention — The intervention is based on the social cognitive theory and the transtheoretical model. There are two principle components, the individual consultation and the small group PA activities. In the individual consultation, assessment of current stage of readiness for PA will be performed first. Then, individualized, stage-matched feedback will be sent to the participants. Small group PA activities will be held every 2 weeks in order to increase learning opportunity by peer interaction, make exercise fun, and introduce a role model.
  Arms: Exercise and physical activity

SUMMARY:
The purpose of this study is to investigate the effects of a 6-month physical activity intervention program on mobility and participation after the termination of a 6-week functional strengthening program for school-age children with spastic diplegia cerebral palsy. The primary outcomes are gross motor function, participation, and physical activity behavior.

ELIGIBILITY:
Inclusion Criteria:

* children with spastic diplegia, aged 6 to 12 year-old, and Gross Motor Function Classification System (GMFCS) level between I to III
* able to stand up from a chair independently and maintain standing for more than 2 seconds without falling
* able to answer questionnaire designed for school-age children
* able to follow verbal instructions

Exclusion Criteria:

* have orthopedic surgery, selective dorsal rhizotomy, or use of a baclofen pump within 6 months
* have orthopedic problems or other medical conditions preventing the child from joining the resistance exercise program, such as obvious LE joint contractures, uncontrolled epilepsy, or cardiopulmonary problems
* hearing loss or using hearing aid

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure | 1.5 months

SECONDARY OUTCOMES:
One-repetition maximum of loaded sit-to-stand | 1.5 months
Gait speed | Week 0, 6, 12, 18, 24, 36, 42, 48, 72
1-minute walk test | 1.5 months
School Function Assessment | 3 months
Pediatric Evaluation of Disability Inventory | 1.5 months
Physical activity status by International Physical Activity Questionnaire and accelerometer | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hua-Fang Liao, MS, Study Chair — Institute of Physical Therapy, National Taiwan University
Locations (1):
- Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan

REFERENCES:
- [Background] Liao HF, Liu YC, Liu WY, Lin YT. Effectiveness of loaded sit-to-stand resistance exercise for children with mild spastic diplegia: a randomized clinical trial. Arch Phys Med Rehabil. 2007 Jan;88(1):25-31. doi: 10.1016/j.apmr.2006.10.006. PMID 17207671